CLINICAL TRIAL: NCT04760301
Title: Local Tranexamic Acid During Vaginal Hysterectomy to Reduce Blood Loss
Brief Title: Local Tranexamic Acid During Vaginal Hysteractomy to Reduce Blood Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yair Daykan, Principal Investigator, Meir Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 0354-19-MMC
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- local tranexamic acid injection to cervix (Experimental): 1 gr of Tranexamic acid diluted in 10 ml saline
  Interventions: Drug: local tranexamic acid injection
- local normal saline injection to cervix (Placebo Comparator): 20 ml of saline
  Interventions: Other: local normal saline injection to cervix

INTERVENTIONS:
Drug: local tranexamic acid injection — local tranexamic acid injection to cervix- 1 g tranexamic acid diluted in 10 ml saline
  Other Names: Hexakapron
  Arms: local tranexamic acid injection to cervix
Other: local normal saline injection to cervix — local normal saline injection to the cervix- 20 ml saline
  Arms: local normal saline injection to cervix

SUMMARY:
Assessing the efficiency of Prophylactic use of local tranexamic acid during vaginal hysterectomy to reduce blood loss during operation

DETAILED DESCRIPTION:
This randomized control trial will investigate whether local tranexamic acid is efficient for decreasing bleeding during vaginal hysterectomy.

The investigators will randomize local placebo (saline) vs. local 1 gr tranexamic acid; local 1gr tranexamic acid diluted in 10 ml saline and local 10 ml saline at the beginning of surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20-90 years old female patients going through vaginal hysterctomy

Exclusion Criteria:

* massive bleeding during operation due to major vessles injury
* known coagulopathies
* sensitivity to tranexamic acid
* medical need in tranexamic acid administration during operation due to bleeding

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blood loss during operation - measure in ml | End of surgery
  At the end of the surgery, surgeon will measure the blood in the suction can

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba, Israel
  - Meir medical center, Kfar Saba

IPD SHARING:
Plan to Share IPD: Undecided